CLINICAL TRIAL: NCT00570687
Title: A Study Comparing Subcutaneous Rapid Acting Insulin and One Formulation of Inhaled Insulin in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-118
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Inhaled Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (1):
- 1 (Experimental): Technosphere Insulin
  Interventions: Drug: Technosphere Insulin

INTERVENTIONS:
Drug: Technosphere Insulin — Inhalation 15U/30U

SUMMARY:
The original protocol was a randomized, open-label, 3-way cross-over study with 9 scheduled visits. The visits comprised an initial screening visit, 3 treatment visits for the meal challenge followed by a 2-6-week blood-loss recovery period, an interim safety visit, 3 sequential visits for the glucose clamp, and a final close-out visit.

Protocol Amendment 1 was a randomized, open-label, 2-way cross-over study with 7 visits for each completed subject. The visits comprise an initial screening visit, 2 treatment visits for the meal challenge followed by a 2-6-week blood-loss recovery period, an interim safety visit, 2 sequential visits for the glucose clamp, and a final close-out visit.

For both the original protocol and Protocol Amendment 1, subjects were hospitalized in the clinical unit for all procedures.

DETAILED DESCRIPTION:
The original protocol was a randomized, open-label, 3-way cross-over study with 9 scheduled visits. The visits comprised an initial screening visit, 3 treatment visits for the meal challenge followed by a 2-6-week blood-loss recovery period, an interim safety visit, 3 sequential visits for the glucose clamp, and a final close-out visit.

After review of the meal challenge data from the Original Protocol design, it became apparent that the TI Inhalation Powder, insulin lispro, and Exubera doses were not well matched, and resulted in significantly higher insulin exposure following insulin lispro than the two inhaled treatments. All meal challenge visits were completed for the 18 subjects enrolled. However, the glucose clamp visits were discontinued since it was discovered that a direct comparison between the treatments was not possible.

The protocol was amended (Amendment 1) to ensure that the insulin exposures between TI Inhalation Powder and insulin lispro were more suited (increased the TI Inhalation Powder doses and decreased the insulin lispro dose). An Exubera arm was not included in Amendment 1 due to the market removal of this product.

Protocol Amendment 1 was a randomized, open-label, 2-way cross-over study with 7 visits for each completed subject. The visits comprise an initial screening visit, 2 treatment visits for the meal challenge followed by a 2-6-week blood-loss recovery period, an interim safety visit, 2 sequential visits for the glucose clamp, and a final close-out visit.

For both the original protocol and Protocol Amendment 1, subjects were hospitalized in the clinical unit for all procedures.

ELIGIBILITY:
Inclusion Criteria:

* Receiving diabetes treatment with insulin for a minimum of 3 months
* Body Mass Index (BMI) of ≤ 34 kg/m2 and ≥ 25 kg/m2
* HbA1c ≤ 8.5% based upon results from a central laboratory
* Non-smoking Males and females ≥ 18 and ≤ 70 years of age
* A clinical diagnosis of type 2 diabetes mellitus for ≥ 12 months

Exclusion Criteria:

* Total daily insulin requirement of ≥ 1.2 U/kg body weight
* Use of Symlin® (pramlintide acetate) and/or Byetta® (exenatide) within the preceding 8 weeks
* Two or more severe hypoglycemic episodes within 6 months of screening
* Any hospitalization or emergency room visit due to poor diabetic control within 6 months of Screening
* Severe complications of diabetes
* Previous exposure to any inhaled insulin product
* Currently using an insulin delivery pump
* Allergy or known hypersensitivity to insulin or to any of the drugs to be used in the trial
* Any clinically important pulmonary disease, confirmed by documented history, pulmonary function testing, or radiologic findings
* Chronic use of systemic steroids
* Inability to perform PFT maneuvers to meet the recommended American Thoracic Society (ATS) standards of acceptability and repeatability
* Significant improvement in spirometry following bronchodilation
* Active respiratory infection
* Seizure disorder
* Significant cardiovascular dysfunction and/or history within 3 months of Screening
* Uncontrolled hypertension with a systolic blood pressure of >160 mm Hg and/or diastolic blood pressure > 95 mm Hg at screening, despite pharmacologic treatment
* Clinical nephrotic syndrome or renal dysfunction or disease
* Cancer (other than an excised cutaneous basal cell carcinoma) within the past 5 years or any history of lung neoplasms
* History of active viral and/or cirrhotic hepatic disease and/or abnormal liver enzymes
* Active infection eg, Human Immunodeficiency Virus (HIV), Hepatitis, or history of severe infection within 30 days of Screening
* Anemia
* A previous diagnosis of systemic autoimmune or collagen vascular disease requiring prior or current treatment with systemic corticosteroids, cytotoxic drugs or penicillamine
* Any concurrent illness, other than diabetes mellitus not controlled by a stable therapeutic regime
* Current or previous chemotherapy or radiation therapy that may result in pulmonary toxicity
* Clinically significant abnormalities on screening laboratory evaluation
* Female subjects who are pregnant, lactating or planning to become pregnant during the clinical trial period
* Female subjects of childbearing potential (defined as pre-menopausal and not surgically sterilized or post-menopausal for less than 2 years) not practicing adequate birth control.
* Current drug or alcohol abuse, or a history of drug or alcohol abuse, that, in the opinion of the PI, would not make the subject a suitable candidate for participation in the clinical trial
* Exposure to any investigational medications or devices within the previous 30 days prior to trial entry or participation in another clinical trial during this trial
* Unable and/or unlikely to comprehend and/or follow the trial protocol
* Concurrent medical or major psychiatric condition which, in the opinion of the PI, makes the subject unsuitable for the clinical trial, or could limit the validity of the informed consent and/or impair the subject's ability to participate in the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Rave, MD, Principal Investigator — Profil Institute for Metabolic Research
Locations (1):
- Profil Institute for Metabolic Research, Neuss, GER, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single-center study was conducted at:
  Profil Institut fur Stoffwechselforschung GmbH Hellersbergstrasse 9 D-41460 Neuss, Germany Principal Investigator: Dr. Klaus Rave
  First subjects first visit: 20 September 2007 Last subject last visit: 30 January 2009
Pre-assignment Details: This randomized, open-label crossover study was conducted in 2 phases: original protocol (TI 45 U, Exubera 4mg and Lispro 12 U) and amendment 1 (TI 60U or TI 90 U, and Lispro 10 U). Both original protocol and amendment 1 had screening visits, meal challenge and glucose clamp visits (with a blood-loss recovery period between them) and final visits.
Groups:
- Amendment 1: TI 60 U Then Insulin Lispro 10 U: 60 U of Technosphere Insulin (TI) administered via inhalation using MedTone inhaler, followed by 10 U subcutaneously administered insulin lispro
- Amendment 1: 10 U Insulin Lispro Then 60 U TI: 10 U subcutaneously administered insulin lispro, followed by 60 U of Technosphere Insulin (TI) administered via inhalation using MedTone inhaler
- Amendment 1: TI 90 U Then 10 U Insulin Lispro: 90 U of Technosphere Insulin (TI) administered via inhalation using MedTone inhaler, followed by 10 U subcutaneously administered insulin lispro
- Amendment 1: 10 U Insulin Lispro Then 90 U TI: 10 U subcutaneously administered insulin lispro, followed by 90 U of Technosphere Insulin (TI) administered via inhalation using MedTone inhaler
- Original Protocol: TI to Insulin Lispro to Exubera: 45 U of Technosphere Insulin (TI) administered via inhalation using MedTone inhaler, followed by 12 U of subcutaneously administered insulin lispro, and then 4 mg of Exubera administered via inhalation
- Original Protocol: TI to Exubera to Insulin Lispro: 45 U of Technosphere Insulin (TI) administered via inhalation using MedTone inhaler, followed by 4 mg of Exubera administered via inhalation, and then 12 U of subcutaneously administered insulin lispro
- Original Protocol: Exubera to Insulin Lispro to TI: 4 mg of Exubera administered via inhalation, followed by 12 U of subcutaneously administered insulin lispro,and then 45 U of Technosphere Insulin (TI) administered via inhalation using MedTone inhaler
- Original Protocol: Exubera to TI to Insulin Lispro: 4 mg of Exubera administered via inhalation, followed by 45 U of Technosphere Insulin (TI) administered via inhalation using MedTone inhaler,. and then 12 U of subcutaneously administered insulin lispro
- Original Protocol: Insulin Lispro to TI to Exubera: 12 U of subcutaneously administered insulin lispro, followed by 45 U of Technosphere Insulin (TI) administered via inhalation using MedTone inhaler, and then 4 mg of Exubera administered via inhalation
- Original Protocol: Insulin Lispro to Exubera to TI: 12 U of subcutaneously administered insulin lispro, followed by 4 mg of Exubera administered via inhalation, and then 45 U of Technosphere Insulin (TI) administered via inhalation using MedTone inhaler
Period: Meal Challenge 1 (1 Day) - Orig Protocol
Arm/Group | Amendment 1: TI 60 U Then Insulin Lispro 10 U | Amendment 1: 10 U Insulin Lispro Then 60 U TI | Amendment 1: TI 90 U Then 10 U Insulin Lispro | Amendment 1: 10 U Insulin Lispro Then 90 U TI | Original Protocol: TI to Insulin Lispro to Exubera | Original Protocol: TI to Exubera to Insulin Lispro | Original Protocol: Exubera to Insulin Lispro to TI | Original Protocol: Exubera to TI to Insulin Lispro | Original Protocol: Insulin Lispro to TI to Exubera | Original Protocol: Insulin Lispro to Exubera to TI
Started | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 1 (7-21 Days) - Orig Protocol
Arm/Group | Amendment 1: TI 60 U Then Insulin Lispro 10 U | Amendment 1: 10 U Insulin Lispro Then 60 U TI | Amendment 1: TI 90 U Then 10 U Insulin Lispro | Amendment 1: 10 U Insulin Lispro Then 90 U TI | Original Protocol: TI to Insulin Lispro to Exubera | Original Protocol: TI to Exubera to Insulin Lispro | Original Protocol: Exubera to Insulin Lispro to TI | Original Protocol: Exubera to TI to Insulin Lispro | Original Protocol: Insulin Lispro to TI to Exubera | Original Protocol: Insulin Lispro to Exubera to TI
Started | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Meal Challenge 2 (1 Day) - Orig Protocol
Arm/Group | Amendment 1: TI 60 U Then Insulin Lispro 10 U | Amendment 1: 10 U Insulin Lispro Then 60 U TI | Amendment 1: TI 90 U Then 10 U Insulin Lispro | Amendment 1: 10 U Insulin Lispro Then 90 U TI | Original Protocol: TI to Insulin Lispro to Exubera | Original Protocol: TI to Exubera to Insulin Lispro | Original Protocol: Exubera to Insulin Lispro to TI | Original Protocol: Exubera to TI to Insulin Lispro | Original Protocol: Insulin Lispro to TI to Exubera | Original Protocol: Insulin Lispro to Exubera to TI
Started | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 2 (7-21 Days) - Orig Protocol
Arm/Group | Amendment 1: TI 60 U Then Insulin Lispro 10 U | Amendment 1: 10 U Insulin Lispro Then 60 U TI | Amendment 1: TI 90 U Then 10 U Insulin Lispro | Amendment 1: 10 U Insulin Lispro Then 90 U TI | Original Protocol: TI to Insulin Lispro to Exubera | Original Protocol: TI to Exubera to Insulin Lispro | Original Protocol: Exubera to Insulin Lispro to TI | Original Protocol: Exubera to TI to Insulin Lispro | Original Protocol: Insulin Lispro to TI to Exubera | Original Protocol: Insulin Lispro to Exubera to TI
Started | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Meal Challenge 3 (1 Day) - Orig Protocol
Arm/Group | Amendment 1: TI 60 U Then Insulin Lispro 10 U | Amendment 1: 10 U Insulin Lispro Then 60 U TI | Amendment 1: TI 90 U Then 10 U Insulin Lispro | Amendment 1: 10 U Insulin Lispro Then 90 U TI | Original Protocol: TI to Insulin Lispro to Exubera | Original Protocol: TI to Exubera to Insulin Lispro | Original Protocol: Exubera to Insulin Lispro to TI | Original Protocol: Exubera to TI to Insulin Lispro | Original Protocol: Insulin Lispro to TI to Exubera | Original Protocol: Insulin Lispro to Exubera to TI
Started | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 3 (7-21 Days) - Orig Protocol
Arm/Group | Amendment 1: TI 60 U Then Insulin Lispro 10 U | Amendment 1: 10 U Insulin Lispro Then 60 U TI | Amendment 1: TI 90 U Then 10 U Insulin Lispro | Amendment 1: 10 U Insulin Lispro Then 90 U TI | Original Protocol: TI to Insulin Lispro to Exubera | Original Protocol: TI to Exubera to Insulin Lispro | Original Protocol: Exubera to Insulin Lispro to TI | Original Protocol: Exubera to TI to Insulin Lispro | Original Protocol: Insulin Lispro to TI to Exubera | Original Protocol: Insulin Lispro to Exubera to TI
Started | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 3 | 2 | 3
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 3 | 2 | 3
Period: Clamp 1 (1 Day) - Orig Protocol
Arm/Group | Amendment 1: TI 60 U Then Insulin Lispro 10 U | Amendment 1: 10 U Insulin Lispro Then 60 U TI | Amendment 1: TI 90 U Then 10 U Insulin Lispro | Amendment 1: 10 U Insulin Lispro Then 90 U TI | Original Protocol: TI to Insulin Lispro to Exubera | Original Protocol: TI to Exubera to Insulin Lispro | Original Protocol: Exubera to Insulin Lispro to TI | Original Protocol: Exubera to TI to Insulin Lispro | Original Protocol: Insulin Lispro to TI to Exubera | Original Protocol: Insulin Lispro to Exubera to TI
Started | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 4 (7-21 Days) - Orig Protocol
Arm/Group | Amendment 1: TI 60 U Then Insulin Lispro 10 U | Amendment 1: 10 U Insulin Lispro Then 60 U TI | Amendment 1: TI 90 U Then 10 U Insulin Lispro | Amendment 1: 10 U Insulin Lispro Then 90 U TI | Original Protocol: TI to Insulin Lispro to Exubera | Original Protocol: TI to Exubera to Insulin Lispro | Original Protocol: Exubera to Insulin Lispro to TI | Original Protocol: Exubera to TI to Insulin Lispro | Original Protocol: Insulin Lispro to TI to Exubera | Original Protocol: Insulin Lispro to Exubera to TI
Started | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Clamp 2 (1 Day) - Orig Protocol
Arm/Group | Amendment 1: TI 60 U Then Insulin Lispro 10 U | Amendment 1: 10 U Insulin Lispro Then 60 U TI | Amendment 1: TI 90 U Then 10 U Insulin Lispro | Amendment 1: 10 U Insulin Lispro Then 90 U TI | Original Protocol: TI to Insulin Lispro to Exubera | Original Protocol: TI to Exubera to Insulin Lispro | Original Protocol: Exubera to Insulin Lispro to TI | Original Protocol: Exubera to TI to Insulin Lispro | Original Protocol: Insulin Lispro to TI to Exubera | Original Protocol: Insulin Lispro to Exubera to TI
Started | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 5 (7-21 Days) - Orig Protocol
Arm/Group | Amendment 1: TI 60 U Then Insulin Lispro 10 U | Amendment 1: 10 U Insulin Lispro Then 60 U TI | Amendment 1: TI 90 U Then 10 U Insulin Lispro | Amendment 1: 10 U Insulin Lispro Then 90 U TI | Original Protocol: TI to Insulin Lispro to Exubera | Original Protocol: TI to Exubera to Insulin Lispro | Original Protocol: Exubera to Insulin Lispro to TI | Original Protocol: Exubera to TI to Insulin Lispro | Original Protocol: Insulin Lispro to TI to Exubera | Original Protocol: Insulin Lispro to Exubera to TI
Started | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Meal Challenge 1 (1 Day) - Amendment 1
Arm/Group | Amendment 1: TI 60 U Then Insulin Lispro 10 U | Amendment 1: 10 U Insulin Lispro Then 60 U TI | Amendment 1: TI 90 U Then 10 U Insulin Lispro | Amendment 1: 10 U Insulin Lispro Then 90 U TI | Original Protocol: TI to Insulin Lispro to Exubera | Original Protocol: TI to Exubera to Insulin Lispro | Original Protocol: Exubera to Insulin Lispro to TI | Original Protocol: Exubera to TI to Insulin Lispro | Original Protocol: Insulin Lispro to TI to Exubera | Original Protocol: Insulin Lispro to Exubera to TI
Started | 4 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 1 (7-21 Days) - Amendment 1
Arm/Group | Amendment 1: TI 60 U Then Insulin Lispro 10 U | Amendment 1: 10 U Insulin Lispro Then 60 U TI | Amendment 1: TI 90 U Then 10 U Insulin Lispro | Amendment 1: 10 U Insulin Lispro Then 90 U TI | Original Protocol: TI to Insulin Lispro to Exubera | Original Protocol: TI to Exubera to Insulin Lispro | Original Protocol: Exubera to Insulin Lispro to TI | Original Protocol: Exubera to TI to Insulin Lispro | Original Protocol: Insulin Lispro to TI to Exubera | Original Protocol: Insulin Lispro to Exubera to TI
Started | 4 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Meal Challenge 2 (1 Day) - Amendment 1
Arm/Group | Amendment 1: TI 60 U Then Insulin Lispro 10 U | Amendment 1: 10 U Insulin Lispro Then 60 U TI | Amendment 1: TI 90 U Then 10 U Insulin Lispro | Amendment 1: 10 U Insulin Lispro Then 90 U TI | Original Protocol: TI to Insulin Lispro to Exubera | Original Protocol: TI to Exubera to Insulin Lispro | Original Protocol: Exubera to Insulin Lispro to TI | Original Protocol: Exubera to TI to Insulin Lispro | Original Protocol: Insulin Lispro to TI to Exubera | Original Protocol: Insulin Lispro to Exubera to TI
Started | 4 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 2 (8 Weeks) - Amendment 1
Arm/Group | Amendment 1: TI 60 U Then Insulin Lispro 10 U | Amendment 1: 10 U Insulin Lispro Then 60 U TI | Amendment 1: TI 90 U Then 10 U Insulin Lispro | Amendment 1: 10 U Insulin Lispro Then 90 U TI | Original Protocol: TI to Insulin Lispro to Exubera | Original Protocol: TI to Exubera to Insulin Lispro | Original Protocol: Exubera to Insulin Lispro to TI | Original Protocol: Exubera to TI to Insulin Lispro | Original Protocol: Insulin Lispro to TI to Exubera | Original Protocol: Insulin Lispro to Exubera to TI
Started | 4 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Clamp 1 (1 Day) - Amendment 1
Arm/Group | Amendment 1: TI 60 U Then Insulin Lispro 10 U | Amendment 1: 10 U Insulin Lispro Then 60 U TI | Amendment 1: TI 90 U Then 10 U Insulin Lispro | Amendment 1: 10 U Insulin Lispro Then 90 U TI | Original Protocol: TI to Insulin Lispro to Exubera | Original Protocol: TI to Exubera to Insulin Lispro | Original Protocol: Exubera to Insulin Lispro to TI | Original Protocol: Exubera to TI to Insulin Lispro | Original Protocol: Insulin Lispro to TI to Exubera | Original Protocol: Insulin Lispro to Exubera to TI
Started | 4 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 3 (7-21 Days) - Amendment 1
Arm/Group | Amendment 1: TI 60 U Then Insulin Lispro 10 U | Amendment 1: 10 U Insulin Lispro Then 60 U TI | Amendment 1: TI 90 U Then 10 U Insulin Lispro | Amendment 1: 10 U Insulin Lispro Then 90 U TI | Original Protocol: TI to Insulin Lispro to Exubera | Original Protocol: TI to Exubera to Insulin Lispro | Original Protocol: Exubera to Insulin Lispro to TI | Original Protocol: Exubera to TI to Insulin Lispro | Original Protocol: Insulin Lispro to TI to Exubera | Original Protocol: Insulin Lispro to Exubera to TI
Started | 4 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Clamp 2 (1 Day) - Amendment 1
Arm/Group | Amendment 1: TI 60 U Then Insulin Lispro 10 U | Amendment 1: 10 U Insulin Lispro Then 60 U TI | Amendment 1: TI 90 U Then 10 U Insulin Lispro | Amendment 1: 10 U Insulin Lispro Then 90 U TI | Original Protocol: TI to Insulin Lispro to Exubera | Original Protocol: TI to Exubera to Insulin Lispro | Original Protocol: Exubera to Insulin Lispro to TI | Original Protocol: Exubera to TI to Insulin Lispro | Original Protocol: Insulin Lispro to TI to Exubera | Original Protocol: Insulin Lispro to Exubera to TI
Started | 4 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Amendment 1: 2-way crossover study of 60 U or 90 U of Technosphere Insulin Inhalation Powder crossed with 10 U of subcutaneous insulin lispro
- Original Protocol: 3-way crossover study of 45 U of Technosphere Insulin Inhalation Powder, 4 mg of Exubera, and 12 U of subcutaneous insulin lispro
- Total: Total of all reporting groups
Arm/Group | Amendment 1 | Original Protocol | Total
Number analyzed (Participants) | 12 | 18 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (7.6) | 54.9 (6.9) | 55.1 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 9 | 15 | 24

OUTCOME MEASURES:

1. Primary Outcome: Time to Minimum Endogenous Glucose Production (EGP) - Meal Challenge
Description: Time to minimum EGP post dose
Time Frame: 0-480 minutes
Population: Amendment 1: Subjects with type 2 diabetes; all received TI and were crossed over to lispro; 3 subjects in the 90 U TI group had insufficient data. Original protocol:Subjects with type 2 diabetes; all subjects received all doses; EGPmin could not be calculated for 1 subject for Exubera and 2 subjects for the other treatments.
Measure: Median (Full Range); unit: Minutes
Groups:
- Amendment 1 - TI Inhalation Powder 90 U; Amendment 1 - TI Inhalation Powder 60U; Amendment 1 - Insulin Lispro 10 U: 2-way crossover study of 60 U or 90 U of Technosphere Insulin Inhalation Powder crossed with 10 U of subcutaneous insulin lispro
- Original Protocol - TI Inhalation Powder 45 U; Original Protocol - Exubera 4 mg; Original Protocol - Insulin Lispro 12 U: 3-way crossover study of 45 U of Technosphere Insulin Inhalation Powder, 4 mg of Exubera, and 12 U of subcutaneous insulin lispro
Arm/Group | Amendment 1 - TI Inhalation Powder 90 U | Amendment 1 - TI Inhalation Powder 60U | Amendment 1 - Insulin Lispro 10 U | Original Protocol - TI Inhalation Powder 45 U | Original Protocol - Exubera 4 mg | Original Protocol - Insulin Lispro 12 U
Number analyzed (Participants) | 3 | 6 | 12 | 16 | 17 | 16
Minutes | 75.0 [20 to 80] | 75.0 [45 to 310] | 125.0 [80 to 210] | 60 [30 to 460] | 160 [80 to 480] | 130 [50 to 350]

2. Primary Outcome: Minimum EGP - Meal Challenge
Description: Minimum calculated EGP per subject as change from baseline
Time Frame: 0-480 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µmol/kg/min
Arm/Group | Amendment 1 - TI Inhalation Powder 90 U | Amendment 1 - TI Inhalation Powder 60U | Amendment 1 - Insulin Lispro 10 U | Original Protocol - TI Inhalation Powder 45 U | Original Protocol - Exubera 4 mg | Original Protocol - Insulin Lispro 12 U
Number analyzed (Participants) | 3 | 6 | 12 | 16 | 17 | 16
µmol/kg/min | -10.29 (4.394) | -6.92 (1.584) | -7.11 (2.018) | -7.59 (3.015) | -7.86 (2.962) | -7.63 (2.709)

3. Primary Outcome: EGP AOC0-480 - Meal Challenge
Description: EGP area over the curve from 0 to 480 minutes postdose
Time Frame: 0-480 minutes
Population: Amendment 1: Subjects with type 2 diabetes. All subjects crossed over to lispro treatment. Original protocol:Subjects with type 2 diabetes; all subjects received all doses; AOC could not be calculated for 1 subject for Exubera and 2 subjects for the other treatments.
Measure: Mean (Standard Deviation); unit: µmol/kg
Arm/Group | Amendment 1 - TI Inhalation Powder 90 U | Amendment 1 - TI Inhalation Powder 60U | Amendment 1 - Insulin Lispro 10 U | Original Protocol - TI Inhalation Powder 45 U | Original Protocol - Exubera 4 mg | Original Protocol - Insulin Lispro 12 U
Number analyzed (Participants) | 6 | 6 | 12 | 16 | 17 | 16
µmol/kg | 2272.8 (266.2) | 2108.7 (498.3) | 2190.9 (674.5) | 2129.4 (764.4) | 2488.3 (845.1) | 1985.9 (623.5)

ADVERSE EVENTS:
Time Frame: From the time the informed consent was signed to 30 days after the last study visit or study-related procedure
Groups:
- Amendment 1 -TI Inhalation Powder 90 U; Amendment 1 - TI Inhalation Powder 60 U; Amendment 1 - Insulin Lispro 10 U: 2-way crossover study of 60 U or 90 U of Technosphere Insulin Inhalation Powder crossed with 10 U of subcutaneous insulin lispro
Arm/Group | Amendment 1 -TI Inhalation Powder 90 U | Amendment 1 - TI Inhalation Powder 60 U | Amendment 1 - Insulin Lispro 10 U | Original Protocol - TI Inhalation Powder 45 U | Original Protocol - Exubera 4 mg | Original Protocol - Insulin Lispro 12 U
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/12 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 5/6 | 4/6 | 1/12 | 5/18 | 1/18 | 7/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amendment 1 -TI Inhalation Powder 90 U (N=6) | Amendment 1 - TI Inhalation Powder 60 U (N=6) | Amendment 1 - Insulin Lispro 10 U (N=12) | Original Protocol - TI Inhalation Powder 45 U (N=18) | Original Protocol - Exubera 4 mg (N=18) | Original Protocol - Insulin Lispro 12 U (N=18)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (10) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MannKind has right to 1st joint multicenter publication. After 1st publication PI may publish data only if PI submits proposed publication to MNKD for review 60 days prior to publication date. MNKD may remove any confidential information. If a multicenter publication is not submitted 12 months after conclusion, abandonment, or termination of the Study at all sites, or if MNKD confirms there will be no multicenter Study publication, PI may publish the Study results subject to MNKD rights herein.